CLINICAL TRIAL: NCT05868083
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Antitumor Activity of SNC-109 CAR-T Cell Therapy in Subjects With Recurrent Glioblastoma
Brief Title: The Safety and Efficacy of SNC-109 CAR-T Cells Therapy the Recurrent Glioblastoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Simnova Biotechnology Co.,Ltd. (Industry)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNC-109-101
Record Dates: First submitted 2023-04-18; First posted 2023-05-22 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2023-05

CONDITIONS: Recurrent Glioblastoma Multiforme
Keywords: CAR-T; GBM
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SNC-109 CAR-T Cells (Experimental): After the operation and pre-infusion evaluation, SNC-109 CAR-T Cells will be evaluated.
  Interventions: Drug: SNC-109 CAR-T Cells

INTERVENTIONS:
Drug: SNC-109 CAR-T Cells — SNC-109 CAR-T Cells, first dose from 2×104 CAR+ T Cells, treatment follows the operation and the next dose would be deiced by SRC

SUMMARY:
This is a single arm clinical study to estimate the safety, tolerability and pharmacokinetic (PK) characteristics of Chimeric Antigen Receptor-modified T cells (CAR-T) SNC-109 in patients with recurrent glioblastoma (r-GBM) and preliminarily evaluate the effectiveness, the immunogenicity of the product, as well as their correlation between the changes of cytokines from baseline level after cellular infusion.

DETAILED DESCRIPTION:
It is planned to recruit about 16 patients with rGBM subjects. The protocol consists of screening period, Lymphocytes apheresis period, Operation period, pre-infusion evaluation (-2~-1 days), infusion (day 0), infusion observation (day 1-post infusion), and follow-up period (last infusion-720 days). The incidence of dose limitation toxicity (DLT) will be observed within 28 days after the first infusion. Subjects in this study will receive multiple infusions, starting with 2×104 CAR+ T cells/dose in the first subject, and the Safety Review Committee (SRC) will evaluate the subsequent dosing regimen, dose, infusion interval, and number of treatment cycles. Subsequent subjects will be evaluated by the SRC on the basis of available PK and safety data, and the SRC will determine the dosing regimen, dose, infusion interval and number of treatment cycles based on observed evidences.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤70，both sexes;
* Diagnosed with a history of glioblastoma, and the recurrent glioblastoma has confirmed by histological/molecular pathology (including astrocytoma World Health Organization (WHO) Grade 4);
* Karnofsky (KPS) ≥60;
* The estimated survival time is ≥8 weeks;
* Blood pregnancy tests for women of childbearing age are negative;
* The patient himself/herself, and/or his/her legal guardian, agree to participate in the trial and sign the informed consent form.

Exclusion Criteria:

* Known allergies to study drugs or drugs that may be used in the study;
* Severe concurrent diseases in the heart, lungs, liver, or other vital organs;
* Hypertension is poorly controlled or accompanied by hypertensive crisis or hypertensive encephalopathy;
* In addition to the glioblastoma, with other severe central nervous system diseases or complications or aggressive malignancies;
* Long-term use of immunosuppressant drugs, or large doses of steroids;
* Received live or attenuated vaccine or other surgery had no related to GBM within 4 weeks prior to Lymphocytes apheresis;
* Lymphocytes apheresis or cell infusion combined with infection or unexplained fever.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-06-24 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment related adverse everts | Up to 28 days after first infusion
  Incidence of adverse events associated with CAR-T cell transfusion within 28 days of the first infusion, abnormal and clinical significant laboratory results
Cmax of SNC-109 Cell count | within 2 years after first infusion
  SNC-109 cell count maximum (Cmax) in peripheral blood (PB) and cerebrospinal fluid (CSF)
Tmax of SNC-109 Cell count | within 2 years after first infusion
  SNC-109 cell count time to Cmax(Tmax) in peripheral blood (PB) and cerebrospinal fluid (CSF)
AUC of SNC-109 Cell count | within 2 years after first infusion
  SNC-109 cell count area under the curve (AUC) in peripheral blood (PB) and cerebrospinal fluid (CSF)
Cmax of SNC-109 CAR vector copy number | within 2 years after first infusion
  SNC-109 CAR vector copy number (VCN) maximum (Cmax) in peripheral blood (PB) and cerebrospinal fluid (CSF)
Tmax of SNC-109 CAR vector copy number | within 2 years after first infusion
  SNC-109 CAR vector copy number (VCN) time to Cmax(Tmax) in peripheral blood (PB) and cerebrospinal fluid (CSF)
AUC of SNC-109 CAR vector copy number | within 2 years after first infusion
  SNC-109 CAR vector copy number (VCN) area under the curve (AUC) in peripheral blood (PB) and cerebrospinal fluid (CSF)
Other relevant PK parameters | within 2 years after first infusion
  Other relevant PK parameters in peripheral blood (PB) and cerebrospinal fluid (CSF)

SECONDARY OUTCOMES:
Objective response rate (ORR) after infusion | within 2 years after first infusion
  The data of objective response rate (ORR) after infusion
Progression free survival (PFS) after infusion | within 2 years after first infusion
  The data of Progression free survival (PFS) after infusion
Overall survival (OS) after infusion | within 2 years after first infusion
  The data of Overall survival (OS) after infusion
Efficacy assesment for the treatment according to iRANO | within 2 years after first infusion
  Assessment of disease response rates according to the Immunological Response Assessment in Neuro-Oncology (iRANO)
Changes of Cytokines after infusion | within 2 years after first infusion
  Changes of cytokines (such as Interleukin-6, Interleukin-8 etc.) in peripheral blood (PB) and cerebrospinal fluid (CSF) pre-and post- infusion and at each of the main follow-up time points, and the time to recovery
Concentration of Human anti-chimeric antibody (HACA) | within 2 years after first infusion
  Detection of changes in peripheral blood and cerebrospinal fluid Human anti-chimeric antibody (HACA)

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, China